CLINICAL TRIAL: NCT03883503
Title: The Influence of Water and Salt Intake on Copeptin Levels During Moderate Alcohol Consumption - a Pathophysiological Study
Brief Title: The Influence of Water and Salt Intake on Copeptin Levels During Moderate Alcohol Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CASCO
Record Dates: First submitted 2019-03-13; First posted 2019-03-21 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Alcohol Drinking
Keywords: Copeptin; Salt-water homeostasis
MeSH Terms: conditions — Alcohol Drinking; Diabetes Insipidus | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Beer alone (Experimental): Consumption of beer (correlated for weight to reach a blood alcohol concentration of 0.8) during 1 hour. Continues measurement of sodium, osmolality, copeptin, urinary sodium, urinary osmolality over 12 hours.
  Interventions: Other: Beer 5%o
- Beer and water (Active Comparator): Consumption of beer and additional water (correlated for weight to reach a blood alcohol concentration of 0.8, 1/3 of water, 2/3 of beer) during 1 hour. Continues measurement of sodium, osmolality, copeptin, urinary sodium, urinary osmolality over 12 hours.
  Interventions: Other: Beer 8.5%o and water
- Beer and stock (Active Comparator): Consumption of beer and additional stock(correlated for weight to reach a blood alcohol concentration of 0.8, 1/3 of stock, 2/3 of beer) during 1 hour. Continues measurement of sodium, osmolality, copeptin, urinary sodium, urinary osmolality over 12 hours.
  Interventions: Other: Beer 8.5%o and stock
- Water alone (Placebo Comparator): Consumption of water alone (correlated for weight to reach a blood alcohol concentration of 0.8, 1/3 of stock, 2/3 of beer) during 1 hour. Continues measurement of sodium, osmolality, copeptin, urinary sodium, urinary osmolality over 12 hours.
  Interventions: Other: Water

INTERVENTIONS:
Other: Beer 5%o — Weight adjusted beer to reach 0.8 blood alcohol content will be given over the time course of 1 hour to the participants
  Arms: Beer alone
Other: Beer 8.5%o and water — Weight adjusted beer to reach 0.8 blood alcohol content and water will be given over the time course of 1 hour to the participants
  Arms: Beer and water
Other: Beer 8.5%o and stock — Weight adjusted beer to reach 0.8 blood alcohol content and stock will be given over the time course of 1 hour to the participants
  Arms: Beer and stock
Other: Water — Water equivalent to the calculated volume of beer will be given over the time course of 1 hour to the participants
  Arms: Water alone

SUMMARY:
The main interest of this study is to investigate the influence of moderate alcohol consumption (beer) on salt-water homeostasis. Therefore, 10 healthy volunteers will participate in 4 Intervention:

* Beer alone
* Beer and water
* Beer and salt (stock/bouillon)
* Water alone During the study day, copeptin, sodium, osmolality and urinary sodium/osmolality will be measured at 6 timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males

Exclusion Criteria:

* Any acute or chronic illness
* History of alcohol dependency
* Alcohol consumption >2 units/day
* Active nicotine abuse
* Gluten intolerance
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, etc. of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Epileptic seizures within the last year
* BMI <18.5 or ≥25.9kg/m2

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Difference in copeptin levels between the interventions | 30 minutes after intervention
  Difference in copeptin levels (pmol/l) between moderate beer consumption and moderate beer consumption with additional water and sodium (stock/bouillon) intake at timepoint 1.5 hours.

SECONDARY OUTCOMES:
Change in copeptin levels between the interventions throughout the observation period of 12 hours | Observation period of 12 hours
  Change in copeptin Levels (pmol/l) from baseline to time-point 1 hour, 1.5 hours, 2.5 hours, 4 hours, 12 hours after start of the Intervention, comparing the interventions
Change in plasma sodium levels between the interventions throughout the observation period of 12 hours | Observation period of 12 hours
  Change in plasma sodium (mmol/l) from baseline to time-point 1 hour, 1.5 hours, 2.5 hours, 4 hours, 12 hours after start of the intervention, comparing the interventions
Change in urinary sodium levels between the interventions throughout the observation period of 12 hours | Observation period of 12 hours
  Change in urinary sodium (mmol/kg) from baseline to time-point 1 hour, 1.5 hours, 2.5 hours, 4 hours, 12 hours after start of the intervention, comparing the interventions
Change in plasma osmolality levels between the interventions throughout the observation period of 12 hours | Observation period of 12 hours
  Change in plasma osmolality (mmol/kg) levels from baseline to time-point 1 hour, 1.5 hours, 2.5 hours, 4 hours, 12 hours after start of the intervention, comparing the interventions
Change in urinary osmolality levels between the interventions throughout the observation period of 12 hours | Observation period of 12 hours
  Change in urinary osmolality (mmol/kg) levels from baseline to time-point 1 hour, 1.5 hours, 2.5 hours, 4 hours, 12 hours after start of the intervention, comparing the interventions
Change in plasma Glucose levels between the interventions throughout the observation period of 12 hours | Observation period of 12 hours
  Change in plasma glucose (mmol/l) levels from baseline to time-point 1 hour, 1.5 hours, 2.5 hours, 4 hours, 12 hours after start of the intervention, comparing the interventions
Change in biomarkers involved in the sodium-water homeostasis between the interventions throughout the observation period of 12 hours | Observation period of 12 hours
  Change in different biomarkers (e.g., Fibroblast growth factor 21, aldosterone, renin, Interleukin 6, Interleukin 8) from baseline to time-point 1 hour, 1.5 hours, 2.5 hours, 4 hours, 12 hours after start of the intervention, comparing the interventions
Difference in urinary excretion between the interventions throughout the observation period of 12 hours | Observation period of 12 hours
  Amount of total urinary excretion (ml) at time-point 1 hour, 1.5 hours, 2.5 hours, 4 hours and 12 hours after start of the intervention, comparing the interventions
Change in blood alcohol content between the interventions throughout the observation period of 12 hours | Observation period of 12 hours
  Change in blood alcohol content (°/oo) from baseline to time-point 1 hour, 1.5 hours, 2.5 hours, 4 hours and 12 hours after start of the intervention, comparing the interventions
Difference in Response to lottery Experiment before and after the intervention | Directly before and 30 minutes after intervention
  Change in decision making before and after the intervention, comparing the interventions

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No